CLINICAL TRIAL: NCT02089581
Title: An Open-label, Randomised, Crossover, Single-dose, Study in Healthy Subjects to Compare the Pharmacokinetics of Two Formulations of a Strong Pain Killer With a Marketed Reference Product in a Fasted or Fed State
Brief Title: A Study of Whether 2 New Oral Formulations of a Strong Pain Killer Release the Same Amount of Drug Into the Body as the Marketed Medication
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mundipharma Research Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HMX1508; 2013-005523-16 (EudraCT Number)
Record Dates: First submitted 2014-02-20; First posted 2014-03-18 (Estimated); Last update posted 2015-09-28 (Estimated); Status verified 2015-09

CONDITIONS: Pain
Keywords: Healthy Volunteer; Pharmacokinetics; Bioequivalence
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Drug (Active Comparator): MR2XXX
  Interventions: Drug: Active comparator MR2XXX
- MRXXX (Experimental): MRXXX capsule 12 hourly
  Interventions: Drug: MRXXX
- MR1XXX (Experimental): MR1XXX capsule, 12 hourly
  Interventions: Drug: MR1XXX
- Experimental (Experimental): Experimental Fed
  Interventions: Drug: MRXXX and MR1XXX

INTERVENTIONS:
Drug: Active comparator MR2XXX — comparison of two new oral formulations with existing formulation
  Other Names: MR2XXX
  Arms: Drug
Drug: MRXXX — MRXXX
  Other Names: Experimental capsule formulation compared to marketed reference product
  Arms: MRXXX
Drug: MR1XXX
  Arms: MR1XXX
Drug: MRXXX and MR1XXX — MRXXX and MR1XXX in fed and fasted state
  Other Names: MRXXX and MR1XXX in fed and fasted state
  Arms: Experimental

SUMMARY:
To determine whether two new oral formulations of a strong pain killer release the drug into the body in a similar pattern as the already marketed reference capsule formulation with or without food.

DETAILED DESCRIPTION:
Comparisons will be made between two new oral formulations and an existing marketed reference capsule formulation to determine whether the release rates of the products are similar or equivalent in a fed or fasted state. Determination is by measurement of drug concentrations in the blood at serial collection time points pre-dose until 32 hours post-dose, following an administration of a single oral dose. Pharmacokinetics parameters of AUC and Cmax are the primary endpoints.

ELIGIBILITY:
Inclusion Criteria

* Healthy male or female subjects aged 18 to 55 inclusive.
* Female subjects who are sexually active or become sexually active must be willing to use highly effective methods of contraception throughout the study. A highly effective method of birth control is defined as one which results in a low failure rate (i.e. less than 1% per year) when used consistently and correctly such as sterilisation, implants, injectables, combined oral contraceptives, some IUDs (Intrauterine Device), or vasectomised partner.
* Female subjects less than one year post-menopausal must have a negative serum pregnancy test and be non-lactating.
* Female subjects who have been post-menopausal for > 1 year and have elevated serum follicle-stimulating hormone (FSH) or are treated with hormone replacement therapy (HRT).
* Male subjects must be willing to use contraception with their partners throughout the study and for 30 days after completion of the study and agree to inform the Investigator if their partner becomes pregnant during this time.
* Body weight ranging from 55 to 100 kg and a BMI ≥ 18.5 and ≤ 29.9.
* Healthy and free of significant abnormal findings as determined by medical history, physical examination, vital signs, laboratory tests and ECG.
* Willing to eat all the food supplied throughout the study.
* The subject's primary care physician has confirmed within the last 12 months that there is nothing in their medical history that would preclude their enrolment into a clinical study.

Exclusion Criteria

* Any history of drug or alcohol abuse.
* Any history of conditions that might interfere with drug absorption, distribution, metabolism or excretion.
* Use of opioid or opioid antagonist-containing medication in the past 30 days.
* Any history of frequent nausea or vomiting regardless of etiology.
* Any history of seizures or symptomatic head trauma.
* Paralytic ileus, respiratory depression, hypoxia or elevated carbon dioxide levels in the blood.
* Participation in a clinical drug study during the 90 days preceding the initial dose in this study.
* Subjects must not participate in both the pilot and definitive phase or in more than one Cohort.
* Any significant illness during the 4 weeks preceding entry into this study.
* Use of any medication including vitamins, herbal and/or mineral supplements during the 7 days preceding the initial dose or during the course of this study (with the exception of the continued use of HRT and contraceptives). Note: subjects taking oral contraceptives containing CYP3A4 inhibitors such as gestodene should be excluded as this may lead to elevated plasma concentrations.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2014-04; Primary Completion 2014-05 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Assess the pharmacokinetics and potential for bioequivalence of two novel formulations | Up to 32 hours
  Areas under the plasma concentration-time curve calculated to the last measurable concentration (AUCt) will be calculated using the linear trapezoidal method. Where possible, the terminal phase rate constants will be estimated using those points determined to be in the terminal log-linear phase. Half-lives (t1/2Z) will be determined from the ratio of ln 2 to LambdaZ. The areas under the plasma concentration-time curve between the last measured point and infinity will be calculated from the ratio of the final observed plasma concentration (Clast) to LambdaZ. This will be added to the AUCt to yield the area under the plasma concentration-time curve between the time of administration and infinity (AUCINF).
The primary objective of the definitive phase is to assess bioequivalence of one or two experimental capsule formulations | 32 hours
  Areas under the plasma concentration-time curve calculated to the last measurable concentration (AUCt) will be calculated using the linear trapezoidal method. Where possible, the terminal phase rate constants will be estimated using those points determined to be in the terminal log-linear phase. Half-lives (t1/2Z) will be determined from the ratio of ln 2 to LambdaZ. The areas under the plasma concentration-time curve between the last measured point and infinity will be calculated from the ratio of the final observed plasma concentration (Clast) to LambdaZ. This will be added to the AUCt to yield the area under the plasma concentration-time curve between the time of administration and infinity (AUCINF). Drug Concentration Measurements: Pre-dose on the first day of each study period, and at 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 16, 24 and 32 hours after dosing (19 samples per study period).

SECONDARY OUTCOMES:
Assess the safety and tolerability of two experimental formulations of Tablet and Capsule in a fasted and fed state by the collection of adverse events, vital signs, clinical laboratory results and ECGs | Up to 32 hours
  Assess the safety and tolerability of two experimental formulations of Tablet and Capsule in a fasted and fed state by the collection of adverse events, vital signs, clinical laboratory results and ECGs

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Biokinetic, Belfast
  - Belfast